CLINICAL TRIAL: NCT02706678
Title: Efficacy and Safety of a Post-transplantation Switch From Cyclosporin to Tacrolimus Sustained-release Capsules in Renal Transplant Recipients: A Multi-center, Open-label, Uncontrolled Study
Brief Title: Efficacy and Safety Study of the Switch From Cyclosporin to Tacrolimus in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJ309CT-02
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Renal Transplant Recipients
Keywords: FK506; Renal transplant recipients; cyclosporin
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus sustained-release capsule group (Experimental): Oral
  Interventions: Drug: Tacrolimus sustained-release capsule

INTERVENTIONS:
Drug: Tacrolimus sustained-release capsule — Oral
  Other Names: FK506

SUMMARY:
The objective of this study is to evaluate the effects of tacrolimus sustained-release capsules replacing cyclosporin on kidney function of renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, male or female
* 1-5 years after kidney transplantation
* The patient has been accepting cyclosporin-based immunosuppressive therapy for ≥6 months, and the therapeutic regimen has kept stable for at least 4 weeks before inclusion
* The dose of cyclosporin has kept stable for at least 4 weeks before inclusion
* At least one of the cyclosporin-related adverse reactions is present or the answer to the 5th question in the questionnaire is "Yes" at the time of inclusion:
* gingival hyperplasia and treatment requested by the patient
* polytrichia and interventional therapy requested by the patient
* post-transplantation hypertension
* post-transplantation hyperlipemia (total cholesterol>5.7 mmol/L (220 mg/dl))
* Serum creatinine<200 μmol/l ( 2.3 mg/dl)
* A promise is made to take contraceptive measures during the study (women at childbearing ages).

Exclusion Criteria:

* Patients having accepted transplantation of other organs apart from kidney transplantation
* Patients with 24-hour urine protein>2 g
* Patients with SGPT/ALT, SGOT/AST or total bilirubin continually increasing to more than twice the normal value(s)
* Patients with refractory infectious foci
* Patients with serious diarrhea or vomiting, active upper gastrointestinal ulcers or malabsorption
* Patients with serious heart or lung diseases or history of sugar tolerance abnormality or malignant tumors
* Patients allergic to tacrolimus or other basic medications
* Pregnant or lactating women
* Patients having participated in other clinical trials within the previous month
* Other patients who are considered by doctors unsuitable for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-12-29 (Actual); Primary Completion 2012-08-01 (Actual); Study Completion 2012-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in creatinine level | Baseline and Week 24

SECONDARY OUTCOMES:
Change from baseline in creatinine level | Baseline and Weeks 1, 2, 4, 8 and 12
Incidence of rejection reaction after drug use | Up to Week 24
Plasma concentrations of tacrolimus | Weeks 1, 2, 4, 8, 12 and 24
Change from baseline in blood pressure | Baseline and Weeks 1, 2, 4, 8, 12 and 24
  Diastolic pressure and systolic pressure
Change from baseline in blood lipid | Baseline and Weeks 1, 2, 4, 8, 12 and 24
  Total cholesterol, high density lipoprotein, low density lipoprotein, triglyceride
Change from baseline in liver function | Baseline and Weeks 1, 2, 4, 8, 12 and 24
  Aspartate aminotransferase, alanine aminotransferase, bilirubin
Change from baseline in fasting blood glucose | Baseline and Weeks 1, 2, 4, 8, 12 and 24
Change from baseline in gingival hyperplasia | Baseline and Week 24
Change from baseline in polytrichia | Baseline and Week 24
Safety assessed by Adverse Events | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (9):
- China (9):
  - Beijing
  - Changchun
  - Chengdu
  - Guangzhou
  - Nanjing
  - Nanning
  - Shanghai
  - Shenyang
  - Wuhan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=202